CLINICAL TRIAL: NCT00905203
Title: Effects of Different Exercise Training Dose on Exercise Performance and Noninvasively Estimated Muscle Oxygen Extraction in Diabetic Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ying-Tai Wu, School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200811009R
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-06

CONDITIONS: Postmenopausal Diabetes
Keywords: Postmenopausal women; Diabetes; Skin microcirculation; Exercise capacity; Skeletal muscle oxygenation; Dose-response relationship; postmenopausal diabetic women
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): moderate exercise training (three times/ week including one home-based training and two supervised training)
  Interventions: Other: exercise
- 2 (Experimental): intensive exercise training (four times/ week including one home-based training and three supervised training)
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — exercise training

SUMMARY:
The purpose of this study is specifically to investigate (1) the exercising muscle oxygenation response in diabetic postmenopausal women; (2) the dose-response of different physical activity interventions on skeletal muscle oxygenation response; (3) the related mechanisms of training effects.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary postmenopausal women
* Ages 45 to 70 years old

Exclusion Criteria:

* Known cardio-respiratory disease
* Diabetic complication
* Excessive weight change during last year
* Cancer and mental disorders

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
skeletal muscle oxygenation response | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan